CLINICAL TRIAL: NCT06522919
Title: Sequential Immunochemotherapy Treatment with Pembrolizumab Plus Dendritic Cell (DC) Vaccine Followed by Trifluridine/Tipiracil (FTD/TPI) Plus Bevacizumab in Refractory Mismatch-repair-proficient (pMMR) or Microsatellite-stable (MSS) Metastatic Colorectal Cancer (CombiCoR-Vax)
Brief Title: Sequential Immunochemotherapy Treatment with Pembrolizumab Plus Dendritic Cell (DC) Vaccine Followed by Trifluridine/Tipiracil Plus Bevacizumab in Refractory Mismatch-repair-proficient (pMMR) or Microsatellite-stable (MSS) Metastatic Colorectal Cancer
Acronym: CombiCoR-Vax
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST153.09
Record Dates: First submitted 2024-07-09; First posted 2024-07-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer Metastatic; Microsatellite Stable Colorectal Carcinoma; Refractory Mismatch-repair-proficient (pMMR) Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Vaccines

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label, multicenter phase 2 clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sequential immunochemotherapy with Pembrolizumab plus DC Vaccine, followed by FTD/TPI + Bevacizumab (Experimental): Induction phase: In the immunological induction phase patients will be given DCs intradermally every week for up to 4 doses and then a further administration after 3 weeks and Pembrolizumab 200 mg IV q3w for up to 3 cycle.
  Maintenance phase: patients will receive FTD/TPI combined with Bevacizumab.Treatment with FTD/TPI and Bevacizumab will start regardless of the response obtained with the induction combo immunotherapy, and will continue until confirmed disease progression, unacceptable toxicity or withdrawal of the consent by the patient, whichever occurs first.
  Interventions: Biological: Autologous Dendritic Cell (DC) Vaccine

INTERVENTIONS:
Biological: Autologous Dendritic Cell (DC) Vaccine — Induction combo immunotherapy (Pembrolizumab plus DC Vaccine) followed by a maintenance chemotherapy (FTD/TPI plus Bevacizumab) in patients with refractory MSS/pMMR metastatic colorectal cancer.

SUMMARY:
Single-arm, open-label, multicenter phase 2 clinical trial evaluating the clinical and the immunological activity of an innovative strategy with an induction combo immunotherapy (Pembrolizumab plus DC Vaccine) followed by a maintenance chemotherapy (FTD/TPI plus Bevacizumab) in patients with refractory MSS/pMMR metastatic colorectal cancer.

DETAILED DESCRIPTION:
Metastatic colorectal cancer (mCRC) remains an incurable disease characterized by a poor prognosis. Recently, in the global phase 3 SUNLIGHT (NCT04737187) study, adding Bevacizumab to Trifluridine/Tipiracil (FTD/TPI) in the treatment of refractory mCRC significantly improved overall survival. Therefore, this combination regimen is going to become the new standard of care for refractory mCRC. Immune checkpoint inhibitors (ICIs), including Pembrolizumab, have shown excellent results in MSI-H or dMMR mCRC, and recent trials evaluating both concomitant and sequential chemoimmunotherapy in MSS/pMMR mCRC (in particular ATEZOTRIBE and MAYA trials), have shown promising results. Since 2001, we have treated more than 80 advanced melanoma patients with a tumor lysate loaded autologous DC vaccine, observing a clinical benefit of 54.1% and, more importantly, an ORR of 63.6% to subsequent chemotherapy, suggesting that immunotherapy might improve the activity of sequential chemotherapy. Moreover, our team has recently concluded the first step of 2 ongoing clinical studies with DC vaccine administration, in radically resected mCRC and metastatic mesothelioma patients - showing that the vaccine was safe and promoted immunological responses that allowed it to continue with patients enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent.
* Histologically confirmed pMMR or MSS mCRC
* Male or female, aged ≥ 18 years
* Life expectancy greater than 12 weeks
* ECOG performance status <2
* Patient suitable for the collection of biological material from leukapheresis: negative serological tests (HIV, HBV, HCV, Treponema pallidum); normal cardiological parameters (12-lead ECG and echocardiogram); evaluation by transfusionist to exclude possible contraindications to leukapheresis; recovered (grade 1 or less by CTCAE 5.0) from all the adverse events related to previous treatments.Exclusion Criteria:
* Patients must have measurable disease by RECIST v 1.1 criteria on CT (or MRI) scan of the chest, abdomen and pelvis. See section 9.2 and Appendix D for the evaluation of measurable disease.
* Prior treatment with 1-2 chemotherapy regimens in an advanced setting, including (if not contraindicated) fluoropyrimidines, irinotecan, oxaliplatin, an anti-VEGF monoclonal antibody and/or anti-EGFR monoclonal antibody for RAS wild-type tumors.
* Patients must have normal organ and marrow function as defined below:

leukocytes >3,000/μL, absolute neutrophil count >1,500/μL, platelets >100,000/μL, total bilirubin < 1.5 X institutional upper limit of normal (ULN), AST(SGOT)/ALT(SGPT) <2.5 X ULN, creatinine < 1.5 X ULN OR creatinine clearance >30 mL/min/1.73 m2

* The autologous surgical specimen needed for vaccine manufacturing must have been collected and sent to the Somatic Cell Therapy Lab of IRCCS IRST and must fulfill all the acceptance criteria prescribed by the GMP procedures
* Recovery (grade 1 or less by CTCAE 5.0) from all the adverse events related to previous surgery.
* A female participant is eligible to participate if she is not pregnant and not breastfeeding. Female patients of childbearing potential and all male patients must accept and be compliant with a highly effective contraceptive method
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

The participant may not enter the study if ANY of the following apply:

* Prior treatment with FTD/TPI for mCRC
* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Pembrolizumab, FTD/TPI, Bevacizumab or components of the DC vaccine.
* History of congenital or acquired immunodeficiency, including history of organ transplantation.
* Any active inflammatory or autoimmune disease requiring systemic steroids or other immunomodulatory agents
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 5 years (except for previously treated basal cell carcinoma and in situ carcinoma of the uterine cervix).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 2 years
  The primary endpoint is Overall Response Rate (ORR) of chemotherapy, defined as the percentage of patients experiencing partial response (PR) or complete response (CR), according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, after starting the treatment with FTD/TPI plus Bevacizumab.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Measured as the time from the start of the treatment with FTD/TPI plus Bevacizumab to the date of first progression, or the date of death from any cause, or the date of the last restaging in non-progressed patients
Safety evaluation | 2 years
  All adverse events will be recorded during the observation period (i.e. from the day of the first DC vaccine dose administered in the induction phase up to 30 days after the last dose of chemotherapy), will be reported and graded according to NCI CTCAE 5.0.
Overall Survival (OS) | 2 years
  Measured from the start of the induction treatment until the date of death from any cause or the last date on which it was known that the patient was alive.
In vivo immunomonitoring through DTH test: | 2 years
  In vivo immunomonitoring through DTH test: DTH testing will be performed in all patients on day 0 (pre-treatment DTH), after the induction phase (post-combo immuno treatment DTH), after the maintenance phase, at the end of treatment and at disease progression. The diameter of induration/erythema observed after 24 hours is recorded according to the following scale: 0-5 mm grade 1, 6-10 mm grade 2, 11-20 mm grade 3, and > 21 mm grade 4. As DTH reactivity to lower concentrations of the antigen(s) is strictly related to more intense antigen specific immune responses, score results will be normalized against the concentration itself and transformed into a 0-80 scale for analysis purposes. Best results obtained for each patient at any of the posttreatment DTHs, either for tumor homogenate or keyhole limpet hemocyanin (KLH), will be taken into account for data analysis (best normalized score).
Characterization of patient's HLA class I immune response | 2 years
  The typing of the locus A-B-C-DR and DQA/DQB will be performed by the Genetic Laboratory by means of the sequence-specific oligonucleotide probe reverse hybridization (PCR-SSO) method. This information will be used to design patient's HLA restricted peptides for personalized functional in vitro immune assays (such as IFN-γ ELISPOT assay and INF-γ secretion assay), as well as for tetramer-guided peripheral monitoring of the antigen specific response. Moreover, statistical analysis will be conducted to correlate the strength of the recorded immunological response to the full HLA haplotype and the clinical outcome.
Characterization of patient's HLA class II immune response | 2 years
  The typing of the locus A-B-C-DR and DQA/DQB will be performed by the Genetic Laboratory by means of the sequence-specific oligonucleotide probe reverse hybridization (PCR-SSO) method. This information will be used to design patient's HLA restricted peptides for personalized functional in vitro immune assays (such as IFN-γ ELISPOT assay and INF-γ secretion assay), as well as for tetramer-guided peripheral monitoring of the antigen specific response. Moreover, statistical analysis will be conducted to correlate the strength of the recorded immunological response to the full HLA haplotype and the clinical outcome.
Characterization of patient's HLA-restricted immune response | 2 years
  The typing of the locus A-B-C-DR and DQA/DQB will be performed by the Genetic Laboratory by means of the sequence-specific oligonucleotide probe reverse hybridization (PCR-SSO) method. This information will be used to design patient's HLA restricted peptides for personalized functional in vitro immune assays (such as IFN-γ ELISPOT assay and INF-γ secretion assay), as well as for tetramer-guided peripheral monitoring of the antigen specific response. Moreover, statistical analysis will be conducted to correlate the strength of the recorded immunological response to the full HLA haplotype and the clinical outcome.
Definition of the prognostic and predictive role of peripheral immune cell subsets and soluble factors | 2 years
  Definition of the prognostic and predictive role of peripheral immune cell subsets and soluble factors: PBMC samples taken before treatment, during and after treatment will be evaluated by multiparametric flow cytometry to assess abundance of regulatory cell subsets (regulatory T cells and immunosuppressive myeloid cells). Moreover, an automated platform of multianalyte will be applied in longitudinal plasma samples. Results will be analyzed by means of bioinformatics and statistical tools and correlated with all the relevant clinical parameters.
In situ characterization of pMMR mCRC through Next Generation Sequencing analysis | 2 years
  NGS approaches (WES and RNAseq analysis) together with in house available bioinformatics pipeline will be used to score the antigen/neoantigen expression in pre-treatment and, whenever available, post-treatment tissue. Deconvolution methods will be used to enumerate immune cells abundance from transcriptional data. Moreover, expression of other TME-related transcripts will be addressed and correlated to the clinical outcome.
In situ characterization of MSS mCRC through Next Generation Sequencing analysis | 2 years
  NGS approaches (WES and RNAseq analysis) together with in house available bioinformatics pipeline will be used to score the antigen/neoantigen expression in pre-treatment and, whenever available, post-treatment tissue. Deconvolution methods will be used to enumerate immune cells abundance from transcriptional data. Moreover, expression of other TME-related transcripts will be addressed and correlated to the clinical outcome.
In situ protein validation at the single cell level | 2 years
  In situ protein validation at the single cell level: using an in-house-developed multiplex immunohistochemistry (IHC), well-known mCRC antigens (i.e. survivin, EGFR, p53, MUC-1, mesothelin) will be monitored at the tissue level.
Identification of tumor infiltrating immune cell subsets | 2 years
  Tumor infiltrating immune cell subsets will be identified and quantified (i.e. positive cell score and close proximity score). Moreover, the predictive effect of the frequency and the distribution of infiltrating immune cell subsets will be correlated with the patient's clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Passardi, Principal Investigator — IRCCS IRST
Locations (2):
- Italy (2):
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori"-IRST S.r.l., Meldola, Forlì Cesena
  - Pia Fondazione di Culto e Religione Azienda Ospedaliera "Card.G.Panico", Tricase, Lecce

REFERENCES:
- [Derived] Passardi A, Sullo FG, Bittoni A, Matteucci L, De Rosa F, Bulgarelli J, Tazzari M, Petrini M, Scarpi E, Testoni S, Miserocchi A, Tartagni O, Zani C, Iaia ML, Toma I, Viola MG, Mita MT, Tamburini E, Ridolfi L. CombiCoR-Vax trial: study protocol for a phase II, single-arm, multicenter trial of sequential pembrolizumab plus dendritic cell vaccine followed by trifluridine/tipiracil and bevacizumab in refractory microsatellite-stable metastatic colorectal cancer. BMC Cancer. 2025 Nov 22;25(1):1921. doi: 10.1186/s12885-025-15371-7. PMID 41275134